CLINICAL TRIAL: NCT06409715
Title: Addressing Kinesiophobia in Post-Meniscoplasty Patients Through Progressive Muscle Relaxation Training and Acupressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gansu University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Junfang Miao, Principal Investigator, Gansu University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: interventional
Record Dates: First submitted 2024-05-02; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Meniscus Tear
MeSH Terms: interventions — Acupressure; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Progressive Muscle Relaxation Training (PMRT) involves a series of 11 steps, each involving muscle tension for 10 seconds, followed by 5 seconds of relaxation, with each step repeated twice. This method, provided by the Chinese Medical Association Audiovisual Publishing House, starts on the third postoperative day if there are no complications, with two 30-minute sessions daily. After PMRT, patients proceed with an Acupressure protocol. The session begins with 5-10 minutes of kneading around the knee and pinching the quadriceps, followed by lighter kneading around the patella and its periphery. Knee movements are made within pain limits. Acupressure targets points Zusanli(S36), Sanyinjiao (SP6), and Yanglingquan(GB34) with pressure held for 10 seconds when soreness or numbness is felt. Each point is treated in 3-5 cycles during the twice-daily, 5-minute sessions, concluding with palm percussion on the calf to relax muscles.
  Interventions: Other: Enhanced Care with PMRT and Acupressure
- Control group (Experimental): Following recommended protocols from "Arthroscopic Surgery and Sports Rehabilitation Nursing" 26, post-meniscectomy patient care primarily involves vital sign monitoring, positional support, dietary management, pain control, psychological support, functional training, and educational initiatives on health matters.
  Interventions: Other: standard care

INTERVENTIONS:
Other: Enhanced Care with PMRT and Acupressure — Progressive Muscle Relaxation Training (PMRT) is a structured strategy created to reduce psychological and physiological stress by alternating muscle contraction and relaxation.Rooted in traditional Chinese medicine's meridian theory, acupressure employs manipulative techniques on distinct acupoints to induce therapeutic effects 18. Targeting enhanced circulation, pain relief, muscle relaxation, and systemic regulation, acupressure's efficacy as both a preventive and therapeutic modality in complementary and alternative medicine is well-established
  Arms: Experimental group
Other: standard care — vital sign monitoring, positional support, dietary management, pain control, psychological support, functional training, and educational initiatives on health matters.
  Arms: Control group

SUMMARY:
The objective of this clinical trial is to determine whether progressive muscle relaxation training and acupressure can reduce kinesiophobia (fear of movement) in patients recovering from meniscoplasty surgery. The study will also monitor the safety of these non-pharmacological interventions. The main questions the trial aims to answer are:

Does the combination of progressive muscle relaxation training and acupressure decrease kinesiophobia in post-meniscoplasty patients? What are the other benefits, if any, of these interventions in terms of pain management and functional mobility? Are there any negative effects associated with these treatments?

Participants in the study will:

Receive progressive muscle relaxation training and acupressure or a placebo control treatment for a duration of 3 months.

Visit the clinic once every month for evaluation and follow-up treatments. Keep a journal recording their fear of movement levels, pain levels, and mobility status.

DETAILED DESCRIPTION:
This study received approval from the Ethics Committee of a tertiary class A hospital in Lanzhou, ID 202159. The research period extended from December 2021 to February 2023. Subjects comprised patients who developed kinesiophobia following meniscus shaping surgery within the Sports Medicine Department of the aforementioned hospital in Lanzhou.

ELIGIBILITY:
Inclusion Criteria:

* Patients confirmed with meniscal damage as per established diagnostic guidelines and subjected to meniscus sculpting surgery
* Individuals post-meniscus surgery exhibiting a Tampa Scale of Kinesiophobia (TSK) score exceeding 37 points
* First-time patients receiving unilateral meniscal surgery
* Exclusive employment of the meniscus sculpting surgical procedure
* Participation were entirely voluntary for all research participants

Exclusion Criteria:

* Patients with compromised consciousness or communicative impairments
* Individuals with a history or presence of post-surgical lower limb thrombosis, resulting in activity limitation
* Patients enduring deformities in the hip or ankle joints
* Those previously engaged in analogous research endeavors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
TSK | Data from TSK were gathered within two days post-operation, on the first day after intervention (i.e., the third postoperative day), the fifth day (i.e., the seventh postoperative day), and on the day of discharge(up to 14 days).
  The Tampa Scale for Kinesiophobia (TSK) The TSK assesses fear of movement/(re)injury and ranges from 17 to 68, indicating the degree of fear; higher scores denote increased apprehension. It has a Cronbach's alpha of 0.70-0.92 and a test-retest reliability above 0.80 28, 29. The Chinese version of TSK was cross-culturally adapted and validated by Wei et al.displaying good reliability (Cronbach's alpha: 0.74) and validity (test-retest reliability: 0.86).
VAS | Data from VAS were gathered within two days post-operation, on the first day after intervention (i.e., the third postoperative day), the fifth day (i.e., the seventh postoperative day), and on the day of discharge(up to 14 days).
  Visual Analogue Scale（VAS） Pain levels were quantified using VAS, which rates pain intensity on a 100 mm line ranging from 0 (no pain) to 10 (severe pain). The VAS is widely deemed a credible and efficacious pain rating tool 31.
KSS | This scoring was performed on the day of patient discharge(up to 14 days).
  American knee society score（KSS ） The KSS scores knee functionality in two domains: self-reported symptoms, signs, and a functional component reflecting walking and stair climbing abilities. Higher scores represent more optimal knee function and mobility capacities. Each KSS domain is rated from 0 to 100 and can be considered individually or collectively.

CONTACTS AND LOCATIONS:
Overall Officials: rui xu, Principal Investigator — Gansu University of Chinese Medicine
Locations (1):
- Chengguanqu, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu R, Miao J, Gong Y, Jia H, Wu H, Wang W, Wang H, Dong M, Zhang Y. A Randomized, Double-Blind, Parallel-Controlled Trial: Addressing Kinesiophobia in Post-Meniscoplasty Patients Through Progressive Muscle Relaxation Training and Acupressure. Pain Res Manag. 2025 Mar 31;2025:1270985. doi: 10.1155/prm/1270985. eCollection 2025. PMID 40201731